CLINICAL TRIAL: NCT04543786
Title: Spinal Excitability Changes and Transcutaneous Spinal Cord Stimulation in Lower Limb Amputees
Brief Title: Neuromodulation in Lower Limb Amputees
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Medical University of South Carolina (Other); Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Lee Fisher, PhD, PhD, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY20060101; P2CHD086844 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-09-10 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: Amputation; Phantom Limb Pain; Hoffman's Reflex
Keywords: Electromyography; Electrical Stimulation; Transcutaneous Spinal Cord Stimulation; Posterior Root-Muscle Reflex
MeSH Terms: conditions — Phantom Limb; Reflex, Abnormal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous spinal cord stimulation (Experimental): Transcutaneous spinal cord stimulation on lower back for 30-60 minutes for 5 consecutive days.
  Interventions: Device: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulation — Neuromodulation with transcutaneous spinal cord stimulation applied on lower back adjacent to spine for 30-60 minutes for 5 consecutive days.

SUMMARY:
The goal of this study is to investigate the role of transcutaneous spinal cord stimulation on spinal cord excitability in lower limb amputees. In this study, the investigators will quantify the spinal cord excitability determined by 1) reflexes and electromyography, and 2) phantom limb pain using self-reported pain assessments. The investigators will assess these measures of spinal excitability in lower limb amputees before and after transcutaneous spinal cord stimulation.

DETAILED DESCRIPTION:
The overall goal of this work is to investigate the changes in the spinal cord resulting from limb amputation. Limb amputation results in an extreme form of peripheral nerve injury. Damage to peripheral nerves, such as with neuropathy, crush injuries, nerve transection, or limb amputation often results in chronic pain, which may be associated with altered excitability of spinal sensorimotor pathways. These spinal pathways become hyperexcitable due to a lack of sensory input, which causes tonic disinhibition of descending circuits and spontaneous activity in the dorsal root ganglia (DRG). Spinal excitability can be measured using the H-reflex, in which electrical stimulation of muscle spindle Ia afferents activates spinal motoneurons via the myotatic reflex, as well as the posterior root-muscle (PRM) reflex, which is elicited by transcutaneous stimulation over the dorsal roots and is considered to be half of the H-reflex, excluding the peripheral primary afferents, but with multiple root activation. Spinal excitability has not been measured in amputees but may offer a potential biomarker for PLP. Neuromodulation may restore normal spinal excitability and reduce PLP, thus offering the potential to improve the quality of life in individuals with a lower limb amputation. The results of this study will provide the foundation for future development of a neuroprosthesis to restore spinal excitability and reduce PLP in individuals with a lower limb amputation. Subjects will undergo 5 testing and stimulation sessions in 1 week. An additional 3 days of recording sessions may be necessary if a phantom limb pain episode does not occur during normal testing days.

Specific Aim 1: Quantify spinal excitability. A lack of sensory input results in spinal hyperexcitability through several pathways including tonic disinhibition of descending circuits and spontaneous activity in the DRG. Spinal cord excitability is directly related to reflex modulation; impaired or enhanced reflex modulation indicates abnormal spinal cord excitability. Spinal cord excitability will be determined in people with a lower limb amputation using the H-reflex and posterior root-muscle (PRM) reflex. The H-reflex is elicited with electrical stimulation of peripheral nerves, exciting muscle spindle Ia afferents projecting to spinal motoneurons via the myotatic reflex. Stimulation of the peripheral nerves also elicits a direct motor (M) wave. The PRM reflex is elicited by electrical stimulation of the posterior roots on the back. It is considered to be half of the H-reflex, excluding the peripheral motor efferents, but activates multiple dorsal roots. Reflex amplitude and latency, threshold, recruitment curves, and rate-dependent depression will be measured and compared to intact controls. The investigators hypothesize that H and PRM reflex hyperexcitability will be present in the residual limb of amputees with PLP. These results will provide insight into the role of limb amputation on spinal cord health and excitability.

Specific Aim 2: Characterize the effects of transcutaneous spinal cord stimulation on spinal cord excitability and phantom limb pain.

Neuromodulation of sensorimotor pathways using transcutaneous electrical nerve stimulation (TENS), dorsal root ganglia stimulation (DRGS), and epidural spinal cord stimulation (eSCS) to reduce phantom limb pain have been explored with mixed results. The most promising methods for pain reduction were DRGS or laterally-placed eSCS, indicating that the DRG and dorsal roots are optimal targets for reducing PLP. However, these methods require surgical implantation of electrodes. Transcutaneous spinal cord stimulation (tSCS) is a non-invasive method for stimulating the dorsal roots in a similar way as eSCS. Through activation of the primary afferents, tSCS may inhibit pain pathways and reduce the hyperexcitability that leads to chronic pain. tSCS in people with spinal cord injury has been shown to restore spinal inhibition and reduce H-reflex hyperexcitability. The investigators hypothesize that tSCS can reduce PLP through modulation of sensorimotor pathways. By comparing the H- and PRM reflex excitability recorded from the residual limb before and after each session of tSCS, a potential mechanism of PLP could be elucidated. H- and PRM reflex modulation, and any differences in the extent of modulation for each, can further inform on the mechanisms of tSCS and how it modulates sensorimotor pathways. The investigators will also quantify the subjects' experience of PLP before and after the 5 days of tSCS and correlate their pain experiences with spinal excitability measures. The investigators will use a visual analog scale and the McGill Pain Questionnaire to assess changes in pain perception. The investigators will also use an algometer to determine changes in local pain threshold.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 21 and 70 years old.
* Participants must have a trans-tibial amputation and phantom limb pain in at least one leg

Exclusion Criteria:

* Participants must not have any serious disease, disorder, or infection (ex. blood or bone disorder or infection) that could affect their ability to participate in this study.
* Female participants of child-bearing potential must not be pregnant or breast feeding, or plan to become pregnant during the course of the study.
* Participants must not have any implanted stimulators or pulse generators
* Participants must not have any implanted metallic devices in their torso and/or legs
* Participants must not have heart disease, including known arrhythmia

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Fisher, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Carnegie Mellon University, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We may share de-identified data with researchers at other centers for the purpose of data analysis and collaboration. We currently do not have a data sharing plan; however, if we decide to share data in the future, we will contact the Office of Sponsored Projects to determine whether an agreement is needed.
  Study sponsors will have access to research data and documents in order to monitor the integrity of the study.
Time Frame: After publication of results. We currently do not have a data sharing plan; however, if we decide to share data in the future, we will contact the Office of Sponsored Projects to determine whether an agreement is needed.
Access Criteria: We currently do not have a data sharing plan; however, if we decide to share data in the future, we will contact the Office of Sponsored Projects to determine whether an agreement is needed.

REFERENCES:
- [Derived] Dalrymple AN, Fisher LE, Weber DJ. A preliminary study exploring the effects of transcutaneous spinal cord stimulation on spinal excitability and phantom limb pain in people with a transtibial amputation. J Neural Eng. 2024 Aug 22;21(4):10.1088/1741-2552/ad6a8d. doi: 10.1088/1741-2552/ad6a8d. PMID 39094627

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcutaneous Spinal Cord Stimulation
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Man | 2
  Gender: Woman | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
H-reflex threshold [Mean (Standard Deviation); unit: mA] — Stimulation amplitude required to evoke of reflex response
  mA | NA (NA) — H-reflexes could not be evoked in any of the participants
PRM threshold [Mean (Standard Deviation); unit: mA] — Stimulation amplitude required to evoke of reflex response
  mA | 59.5 (6.1)
Phantom limb pain score [Mean (Standard Deviation); unit: Score on a Scale] — McGill Pain Questionnaire: minimum = 0, maximum = 78; the higher the pain score, the worse the pain experienced
  Score on a Scale | 34 (7)
Pain pressure threshold [Mean (Standard Deviation); unit: Newton] — Pain Pressure Threshold Test using an algometer: minimum force that induces a painful response
  Newton | 23.84 (13.08)
Pain score [Mean (Standard Deviation); unit: Score on a Scale] — Visual analog scale: minimum = 0, maximum = 10; the higher the score, the greater the pain experienced
  Score on a Scale | 6 (2)
Side of limb amputation [Count of Participants; unit: Participants]
  Left | 2
  Right | 1
Nature of limb amputation [Count of Participants; unit: Participants]
  Trauma | 1
  Diabetic Neuropathy | 1
  Alcohol Neuropathy | 1
Time since amputation [Count of Participants; unit: Participants]
  < 6 months | 1
  >= 5 years | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean H-reflex Threshold
Description: Reflex threshold: stimulation amplitude required to evoke reflex response. The presence of H-reflexes are expected in uninjured individuals.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | NA (NA) — H-reflexes could not be evoked in any of the participants

2. Primary Outcome: Mean H-reflex Threshold
Description: as for outcome 1
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | NA (NA) — H-reflexes could not be evoked in any of the participants

3. Primary Outcome: Mean H-reflex Threshold
Description: as for outcome 1
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | NA (NA) — H-reflexes could not be evoked in any of the participants

4. Primary Outcome: Mean H-reflex Threshold
Description: as for outcome 1
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | NA (NA) — H-reflexes could not be evoked in any of the participants

5. Primary Outcome: Mean PRM Reflex Threshold
Description: Reflex threshold: stimulation amplitude required to evoke reflex response. Thresholds in uninjured people have been reported to be approximately 30 mA.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | 56.7 (4.9)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy. Comparing values at baseline and Day 2; p = 0.0048, ANOVA — Bonferroni post-hoc tests; p < 0.05 was considered significant; One-way; Mean Difference (Final Values) = 2.8

6. Primary Outcome: Mean PRM Reflex Threshold
Description: as for outcome 5
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | 55.8 (5.9)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy. Comparing values at baseline and Day 3; p < 0.001, ANOVA — Bonferroni post-hoc tests; p < 0.05 was considered significant; Mean Difference (Final Values) = 3.72

7. Primary Outcome: Mean PRM Reflex Threshold
Description: as for outcome 5
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | 56.2 (7.6)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy. Comparing values at baseline and Day 4; p < 0.001, ANOVA — Bonferroni post-hoc tests; p < 0.05 was considered significant; Mean Difference (Final Values) = 3.24

8. Primary Outcome: Mean PRM Reflex Threshold
Description: as for outcome 5
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
mA | 38.6 (12.2)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy. Comparing values at baseline and Day 5; p < 0.001, ANOVA — Bonferroni post-hoc tests; p < 0.05 was considered significant; Mean Difference (Final Values) = 20.84

9. Secondary Outcome: Phantom Limb Pain Score
Description: McGill Pain Questionnaire: minimum = 0, maximum = 78, the higher the pain score the greater the pain
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
Score on a Scale | 18.3 (6.8)

10. Secondary Outcome: Pain Pressure Threshold
Description: Pain Pressure Threshold Test using an algometer: minimum force that induces pain, minimum = 0 N, maximum = 444.8 N, a lower threshold indicates hypersensitivity
Time Frame: Day 5
Population: One participant excluded from this analysis due to inconsistent pain medication use on last testing day
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 2
Newton | 50.67 (26.07)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy. Comparing values at baseline and Day 5; p < 0.001, t-test, 2 sided — p < 0.05 was considered significant; paired; Mean Difference (Final Values) = 26.78

11. Secondary Outcome: Pain Score
Description: Visual analog scale: minimum = 0, maximum = 10, the higher the score the greater the pain
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
Score on a Scale | 4.7 (1.5)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy; p = 0.56, ANOVA — p < 0.05 was considered significant; Repeated measures; Mean Difference (Final Values) = 1.3

12. Secondary Outcome: Pain Score
Description: Visual analog scale: minimum = 0, maximum = 10, the higher the score the greater the pain
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
Score on a Scale | 3.7 (3.2)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy; p = 0.56, ANOVA — p < 0.05 was considered significant; Repeated measures; Mean Difference (Final Values) = 2.3

13. Secondary Outcome: Pain Score
Description: Visual analog scale: minimum = 0, maximum = 10, the higher the score the greater the pain
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
Score on a Scale | 4.8 (1.0)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy; p = 0.56, ANOVA — p < 0.05 was considered significant; Repeated measures; Mean Difference (Final Values) = 1.2

14. Secondary Outcome: Pain Score
Description: Visual analog scale: minimum = 0, maximum = 10, the higher the score the greater the pain
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Transcutaneous Spinal Cord Stimulation
Number analyzed (Participants) | 3
Score on a Scale | 4.5 (0.5)
Statistical Analysis 1: Comparison: Transcutaneous Spinal Cord Stimulation; Test type: Other — No comparison was made to another intervention or therapy; p = 0.56, ANOVA — p < 0.05 was considered significant; Repeated measures; Mean Difference (Final Values) = 1.5

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Transcutaneous Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT04543786/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT04543786/ICF_000.pdf